CLINICAL TRIAL: NCT00338793
Title: A Multicenter, Placebo-Controlled, Double-Blind, Randomized Clinical Trial to Evaluate the Efficacy and Safety of Corticosteroids for Treatment of Patients With Tuberculous Pleurisy
Brief Title: Corticosteroids in the Treatment of Tuberculous Pleurisy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangxi Medical University (Other)
Collaborators: National Natural Science Foundation of China (Other Government); Ministry of Education, China (Other Government); Bureau of Science and Technology of Guangxi Province, China (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Shi-TB-01
Record Dates: First submitted 2006-06-19; First posted 2006-06-20 (Estimated); Last update posted 2008-08-26 (Estimated); Status verified 2008-08

CONDITIONS: Tuberculous Pleurisy
Keywords: Tuberculosis;; Pleural effusion;; Corticosteroids.
MeSH Terms: conditions — Tuberculosis, Pleural; Tuberculosis; Pleural Effusion | interventions — Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: prednisolone

SUMMARY:
Tuberculous pleurisy is associated with inflammation and fibrosis. Adjunctive corticosteroids are used for tuberculous pleurisy because their anti-inflammatory effect is thought to minimise pleural reactivity and thereby reduce residual pleural thickening. The purpose is to evaluate the efficacy and safety of oral prednisolone for treatment of adult patients with tuberculous pleurisy.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent;
* Presented with clinical features suggesting pleural tuberculosis;
* Had not previously received treatment or prophylaxis for tuberculosis;
* Had not recently received treatment with glucocorticoids;
* Were not pregnant or breast-feeding.

Exclusion Criteria:

* Failed to complete the screening procedures;
* Were seropositive for HIV
* Tuberculous meningitis;
* Had risk factors for serious steroid-related adverse events (a history of diabetes or positive urine glucose, a history or clinical finding of hypertension, or a history of peptic ulcer disease or mental illness);
* Standard doses of antituberculosis drugs could not be used (as in participants with concurrent liver disease)
* Psychiatric illness;
* Alcoholism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2006-07; Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Death
Presence of pleural thickening
Pulmonary function at completion of treatment
Adverse drug effects

SECONDARY OUTCOMES:
Improvement in clinical symptoms and signs (such as pleuritic chest pain, temperature)
Reabsorption of pleural effusion
Failure rate at the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Huan-Zhong Shi, MD, PhD, Study Chair — Institute of Respiratory Diseases, First Affiliated Hospital, Guangxi Medical University, Nanning 530021, Guangxi, China; Zhan-Cheng Gao, MD, PhD, Principal Investigator — Department of Respiratory Diseases, People's Hospital, Peking University, Beijing, China; Xin Zhou, MD, Principal Investigator — Department of Respiratory Diseases, First Affiliated Hospital, Shanghai Jiaotong University, Shanghai, China
Locations (1):
- Huan-Zhong Shi, Nanning, Guangxi, China